CLINICAL TRIAL: NCT00188747
Title: Comparison of Three Management Strategies for Post Cardiac Surgery Coagulopathy.
Brief Title: Comparison of Three Management Strategies for Post Cardiac Surgery Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Anemia Institute for Research & Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHN REB 05-0054-B; Anemia Institute #04-14
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-04

CONDITIONS: Heart Disease; Coagulopathy
Keywords: Coagulopathy; Cardiac Surgery; Point of Care; Monitoring
MeSH Terms: conditions — Heart Diseases; Hemostatic Disorders | interventions — Point-of-Care Systems

INTERVENTIONS:
Procedure: Thromboelastograph, Point of Care

SUMMARY:
Open-heart surgery frequently results in abnormal clotting, which in turn results in excessive blood loss and the need for transfusion of multiple blood products to patients and leads to adverse outcomes. Prompt identification of any clotting abnormalities after cardiac surgery reduces blood loss and blood product transfusion and may improve outcomes. Currently, however, this monitoring is dependent on standard laboratory-based tests of clotting that have a long turnaround time (30-45 min) and do not measure some important aspect of clotting. There are now other monitoring options that are carried out at patients' bedside, providing results more quickly than standard laboratory tests (within 2-5 minutes for some), and measure more aspects of clotting, providing more information on possible causes of any abnormalities. In this study, we will compare the cost-effectiveness of two of these newer monitoring techniques with standard laboratory-based tests by assigning 150 patients who will be undergoing open-heart surgery to one of the three monitoring techniques (50 patients will be assigned by chance to each group). In each group, an explicit algorithm based on the monitoring technique of that group will be used to guide all transfusion decisions. Between-group differences in number of units of blood products transfused (primary outcome), amount of blood loss, rate of adverse events, and cost of monitoring will be measured. The objective of the study is to determine which of the three methods is most cost-effective in terms of these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years
* no emergent complex cardiac surgery

Exclusion Criteria:

* Isolated CABG
* Single valve surgery
* Pre-existing coagulopathy PTT>50's, INR>1.3
* Severe Thrombocytopenia Platelet <100,000
* Recent Antiplatelet drugs(Plavix within 7 days, Integrilin within 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-06

PRIMARY OUTCOMES:
Units of blood products transfused in the first 24 hours post CPB.

SECONDARY OUTCOMES:
Test cost, chest tube blood loss 24h; blood products in the postoperative period; modifications in transfusion that would have occurred if result from other group's tests were available; length of stay ICU and hospital; incidence of major complications.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada